CLINICAL TRIAL: NCT03677505
Title: Comparison of the KoMAC Videolaryngoscope With the Macintosh Laryngoscope for Double-lumen Intubation
Brief Title: KoMAC Videolaryngoscope for Double-lumen Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-MED-OBS-18-286
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Intubation
Keywords: double lumen intubation; videolaryngoscope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KoMAC group (Experimental): Orotracheal intubation with KoMAC videolaryngoscope
  Interventions: Device: KoMAC videolaryngoscope
- Macintosh group (Active Comparator): Orotracheal intubation with Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: KoMAC videolaryngoscope — Double lumen endotracheal intubation was performed with the KoMAC videolaryngoscope
  Arms: KoMAC group
Device: Macintosh Laryngoscope — Double lumen endotracheal intubation was performed with the Macintosh Laryngoscope
  Arms: Macintosh group

SUMMARY:
KoMAC videolaryngoscope is a portable intubating device with an angulated single-use blade of adjustable size and a liquid crystal display monitor mounted on top of the handle, which is similar in shape to the McGrath videolaryngoscope. The purpose of this study was to evaluate the efficacy of the KoMAC videolaryngoscope for double-lumen intubation regarding intubation time, laryngeal view and ease of intubation, compared to Macintosh laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for thoracic surgery requiring one lung ventilation

Exclusion Criteria:

* predicted difficult airway
* rapid sequence intubation
* cervical injury

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Intubation time | from 2 min after rocuronium injection to completion of intubation (time interval is about 120 seconds)
  Time interval between laryngoscope passing the teeth to the confirming of end tidal CO2

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea